CLINICAL TRIAL: NCT02698488
Title: Embryo Selection by Metabolomic Profiling of Embryo Culture Medium With Mass Spectroscopy as an Adjunct to Morphology: a Randomized Controlled Trial
Brief Title: Embryo Selection by Metabolomic Profiling of Embryo Culture Medium With Mass Spectroscopy as an Adjunct to Morphology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul University (Other)
Collaborators: Acibadem Fulya Hospital (Other); Marmara University (Other)
Responsible Party: Principal Investigator, Ercan Bastu, Associate Professor of Obstetrics and Gynecology, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 201603
Record Dates: First submitted 2016-02-29; First posted 2016-03-03 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Embryo Selection; IVF; Morphology
MeSH Terms: interventions — Mass Spectrometry

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Embryo Selection by Morphology (Active Comparator): Embryos will be morphologically evaluated according to the number and regularity of blastomeres and fragmentation degree. Only embryo culture media of good quality embryos (embryos with ≥6 cells with no fragmentation) will be included in the study
  Interventions: Procedure: Morphology; Procedure: Morphology and Mass Spectroscopy
- Embryo Selection by Morphology and Mass Spectroscopy (Active Comparator): Embryos will be morphologically evaluated according to the number and regularity of blastomeres and fragmentation degree. Only embryo culture media of good quality embryos (embryos with ≥6 cells with no fragmentation) will be included in the study. After dilution, embryo culture media will be analyzed by electrospray ionization quadrupole time-of-flight (ESI-QTOF) MS. The spectra will be collected in the negative ion mode. Abundance of ions in each spectrum will be further analyzed.
  Interventions: Procedure: Morphology; Procedure: Morphology and Mass Spectroscopy

INTERVENTIONS:
Procedure: Morphology
Procedure: Morphology and Mass Spectroscopy

SUMMARY:
Identification of the embryo with the highest potential to implant and establish an ongoing pregnancy is a primary aim in human assisted reproduction. This task is undertaken every day by embryologists worldwide during the treatment of couples that wish to conceive by IVF. The optimal scenario is the transfer of a single embryo which gives rise to a singleton pregnancy. The current limitations in determination of embryos that have the highest implantation potential probably contribute to the low rates of pregnancy during IVF treatments. Hence, since the beginning of IVF, how to improve embryo selection has been a 'hot research topic.' Morphology has been a very obvious parameter to assess embryos as it provides a chance to evaluate them from the oocyte stage all the way to the blastocysts stage. Hence, in the first era of IVF, there were number of studies that evaluated this parameter and associated morphology with IVF success rates. On the other hand, it has been previously stated that the slight increase in pregnancy rates during IVF treatment is mostly likely a result of better practices in laboratory than morphological evaluation. Due to the limitations of morphological evaluation, several researchers have investigated adjunctive non-invasive approaches for the assessment of the embryo, such as the metabolomic profiling.

Recently mass spectroscopic (MS) approaches have been utilized in limited settings. Samples needed minimal preparation; analytical analysis was rapid and large amounts of data was available. Hence, MS might be a promising approach for metabolomic profiling of embryo culture media.

ELIGIBILITY:
Inclusion Criteria:

* any infertility etiology
* good previous response to IVF with ≥1 embryo

Exclusion Criteria

* poor response to IVF previously

Ages: 21 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Clinical Pregnancy | 3 months
  Clinical pregnancy will be defined as the presence of a fetal heartbeat using vaginal ultrasound at 6 weeks of amenorrhoea.

CONTACTS AND LOCATIONS:
Overall Officials: Ercan Bastu, M.D., Principal Investigator — Istanbul University School of Medicine
Locations (1):
- Istanbul University School of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No